CLINICAL TRIAL: NCT04414592
Title: Safety and Effectiveness of Human Umbilical Cord Mesenchymal Stem Cells For the Treatment of Lumbar Disc Degeneration Disease
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells For the Treatment of Lumbar Disc Degeneration Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qiang Fu, Dean of the Minimally Invisive Spine Surgery Department, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QFu
Record Dates: First submitted 2020-05-06; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Lumbar Disc Degeneration; Lumbar Disc Herniation
Keywords: Lumbar Disc Degeneration; Human Umbilical Cord Mesenchymal Stem Cells; Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord Mesenchymal Stem Cells (Experimental): Injection of twenty million human umbilical cord mesenchymal stem cells into the degenerative disc
  Interventions: Other: human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Other: human umbilical cord mesenchymal stem cells — Twenty million human umbilical cord mesenchymal stem cells will be immediately injected into the degenerative discs of such patients who are diagnosed with lumbar disc herniation and operated with full endoscopy lumbar discectomy.

SUMMARY:
This study aims to investigate the safety and efficiency of Human Umbilical Cord Mesenchymal Stem Cells (hUCMSC) for treating lumbar disc degeneration diseases. We hypothesize grafting hUCMSC into the degenerative disc leads to symptoms relief and slow down the progression of disc degeneration.

DETAILED DESCRIPTION:
Lumbar disc herniation causes patients severe lower back pain and radicular pain to decrease the quality of life and lead to great economic burden to patients and society. In recent years, full endoscopic discectomy has been widely used in the treatment of lumbar disc herniation due to its advantages of reduced trauma, enhanced recovery and less cost. However, the reherniation of the residual nucleus pulposus still exist after nerve root decompression. It is urgent to use stem cell and tissue engineering to replace the resection tissue and repair the residual nucleus pulposus for disc resealing. To observe the safety and efficacy of human umbilical cord mesenchymal stem cells (hUCMSCs) in the treatment of lumbar disc degeneration. This clinical trial is aimed to include a single group of 20 patients with lumbar disc herniation. Twenty million hUCMSCs will be injected into the lumbar disc of the enrolled patients in this non-random, self-controlled and single-dose open study design. The patients will be followed up for 3 months, 6 months and 12 months after the injection to evaluate the safety of the patients after grafting hUCMSCs. Additionally, improvement of patients' quality of life will be evaluated using the ODI score, VAS score and SF-36 score. Lumbar disc signals will be also quantified using MRI to demonstrate hUCMSCs transplantation could slow down lumbar disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old;
2. Symptoms with lower back pain and unilateral radicular pain;
3. Failure of conservative treatments including physical therapy, manipulation therapy and non-morphine drug therapy;
4. CT/MRI clearly showing unilateral nucleus pulposus herniation to compress the nerve root;
5. Symptoms and imaging showing unilateral lumbar disc herniation;
6. Imaging showed single-segment lumbar disc herniation;
7. Pfirrmann disc degeneration classification from lumbar MRI: grade I-IV;
8. Segments of lumbar disc herniation: L3-4, L4-5, L5-S1;
9. Unilateral full endoscopic lumbar discectomy;
10. Signing the informed consent;
11. No previous history of spinal surgery.

Exclusion Criteria:

1. Previous history of tumor or spinal infection;
2. Severe coagulation disorders or are taking oral anticoagulants
3. coma or incapacity;
4. MRI contraindications (cardiovascular and cerebrovascular stent implantation history, cardiac pacemaker, biological stimulator, etc.);
5. pregnant;
6. pregnancy or breastfeeding;
7. participated in other clinical trials in the past 30 days;
8. History of stem cell therapy;
9. poor compliance, or inability to properly understand the coordination;
10. received intervertebral disc interventional therapy, such as radiofrequency, laser ablation, protease injection and ozone injection in the past 3 months;
11. Highly allergic constitution or severe allergic history;
12. Severe autoimmune diseases or receiving immunosuppressive therapy;
13. Severe infection or high fever;
14. Shock, failure of vital organs or unstable vital signs;
15. X-ray showing that the stenosis percentage of the degenerative segment was larger than 30% compared to that of the adjacent normal segment.
16. Lumbar disc herniation with calcification;
17. Lumbar disc herniation with Modic Change;
18. Lumbar disc herniation with severe spinal stenosis;
19. Lumbar disc herniation with lumbar spondylolisthesis;
20. Lumbar disc herniation with spinal deformity;
21. psychosocial abnormalities, cognitive impairment, or other physical diseases affecting the research results;
22. Other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Lumbar disc signaling values from magnetic resonance imaging | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in Lumbar disc signaling values from magnetic resonance imaging

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) (0-10 scores, the higher scores mean a worse outcome) | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in Visual Analogue Scale of Lower back pain and leg pain
Oswestry Disability Index(ODI) (0-50 scores, the higher scores mean a worse outcome) | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in Oswestry Disability Index
The Short Form (36) Health survey (SF36) (0-100 scores, the higher scores mean a better outcome) | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in The Short Form (36) Health survey (SF36)
Disc Height Index (DHI) from X ray | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in Disc Height Index
Size of herniated nucleus pulposus from magnetic resonance imaging | Baseline, post-op 3months, post-op 6months, post-op 12months
  Changes from baseline in size of nucleus pulposus from magnetic resonance imaging
Number of participants with treatment-related adverse events by CTCAE v4.0 | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Assessing for worsening of patients' baseline symptoms or functions (will be considered an AE); (also general AE events), particular AE events related to the procedures/treatment. All AEs will be assessed by common terminology criteria for adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Fu, M.D., Principal Investigator — Minimally Invasive Spinal of Shanghai General Hospital
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
All the relative individual participant data (IPD) collected during the trial after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: The researchers associate with disc degeneration and stem cells.

REFERENCES:
- [Background] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Background] Ghiselli G, Wang JC, Bhatia NN, Hsu WK, Dawson EG. Adjacent segment degeneration in the lumbar spine. J Bone Joint Surg Am. 2004 Jul;86(7):1497-503. doi: 10.2106/00004623-200407000-00020. PMID 15252099
- [Background] Chen Z, Zhang L, Dong J, Xie P, Liu B, Wang Q, Chen R, Shu T, Li S, Feng F, Yang B, He L, Yang Y, Liu Z, Pang M, Rong L. Percutaneous Transforaminal Endoscopic Discectomy Versus Microendoscopic Discectomy for Lumbar Disc Herniation: Two-Year Results of a Randomized Controlled Trial. Spine (Phila Pa 1976). 2020 Apr 15;45(8):493-503. doi: 10.1097/BRS.0000000000003314. PMID 31703056
- [Background] Li Z, Lang G, Chen X, Sacks H, Mantzur C, Tropp U, Mader KT, Smallwood TC, Sammon C, Richards RG, Alini M, Grad S. Polyurethane scaffold with in situ swelling capacity for nucleus pulposus replacement. Biomaterials. 2016 Apr;84:196-209. doi: 10.1016/j.biomaterials.2016.01.040. Epub 2016 Jan 21. PMID 26828684
- [Background] Moriguchi Y, Mojica-Santiago J, Grunert P, Pennicooke B, Berlin C, Khair T, Navarro-Ramirez R, Ricart Arbona RJ, Nguyen J, Hartl R, Bonassar LJ. Total disc replacement using tissue-engineered intervertebral discs in the canine cervical spine. PLoS One. 2017 Oct 20;12(10):e0185716. doi: 10.1371/journal.pone.0185716. eCollection 2017. PMID 29053719
- [Background] Benneker LM, Andersson G, Iatridis JC, Sakai D, Hartl R, Ito K, Grad S. Cell therapy for intervertebral disc repair: advancing cell therapy from bench to clinics. Eur Cell Mater. 2014 May 6;27:5-11. doi: 10.22203/ecm.v027sa02. PMID 24802611
- [Background] Sobajima S, Vadala G, Shimer A, Kim JS, Gilbertson LG, Kang JD. Feasibility of a stem cell therapy for intervertebral disc degeneration. Spine J. 2008 Nov-Dec;8(6):888-96. doi: 10.1016/j.spinee.2007.09.011. Epub 2007 Dec 21. PMID 18082460
- [Background] Sakai D, Mochida J, Yamamoto Y, Nomura T, Okuma M, Nishimura K, Nakai T, Ando K, Hotta T. Transplantation of mesenchymal stem cells embedded in Atelocollagen gel to the intervertebral disc: a potential therapeutic model for disc degeneration. Biomaterials. 2003 Sep;24(20):3531-41. doi: 10.1016/s0142-9612(03)00222-9. PMID 12809782
- [Background] Sakai D, Mochida J, Iwashina T, Hiyama A, Omi H, Imai M, Nakai T, Ando K, Hotta T. Regenerative effects of transplanting mesenchymal stem cells embedded in atelocollagen to the degenerated intervertebral disc. Biomaterials. 2006 Jan;27(3):335-45. doi: 10.1016/j.biomaterials.2005.06.038. Epub 2005 Aug 19. PMID 16112726
- [Background] Sakai D, Mochida J, Iwashina T, Watanabe T, Nakai T, Ando K, Hotta T. Differentiation of mesenchymal stem cells transplanted to a rabbit degenerative disc model: potential and limitations for stem cell therapy in disc regeneration. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2379-87. doi: 10.1097/01.brs.0000184365.28481.e3. PMID 16261113
- [Background] Crevensten G, Walsh AJ, Ananthakrishnan D, Page P, Wahba GM, Lotz JC, Berven S. Intervertebral disc cell therapy for regeneration: mesenchymal stem cell implantation in rat intervertebral discs. Ann Biomed Eng. 2004 Mar;32(3):430-4. doi: 10.1023/b:abme.0000017545.84833.7c. PMID 15095817
- [Background] Zhang YG, Guo X, Xu P, Kang LL, Li J. Bone mesenchymal stem cells transplanted into rabbit intervertebral discs can increase proteoglycans. Clin Orthop Relat Res. 2005 Jan;(430):219-26. doi: 10.1097/01.blo.0000146534.31120.cf. PMID 15662327
- [Background] Ho G, Leung VY, Cheung KM, Chan D. Effect of severity of intervertebral disc injury on mesenchymal stem cell-based regeneration. Connect Tissue Res. 2008;49(1):15-21. doi: 10.1080/03008200701818595. PMID 18293174
- [Background] Yi Z, Guanjun T, Lin C, Zifeng P. Effects of Transplantation of hTIMP-1-Expressing Bone Marrow Mesenchymal Stem Cells on the Extracellular Matrix of Degenerative Intervertebral Discs in an In Vivo Rabbit Model. Spine (Phila Pa 1976). 2014 May 15;39(11):E669-E675. doi: 10.1097/BRS.0000000000000316. PMID 24718065
- [Background] Wei A, Tao H, Chung SA, Brisby H, Ma DD, Diwan AD. The fate of transplanted xenogeneic bone marrow-derived stem cells in rat intervertebral discs. J Orthop Res. 2009 Mar;27(3):374-9. doi: 10.1002/jor.20567. PMID 18853431
- [Background] Jeong JH, Jin ES, Min JK, Jeon SR, Park CS, Kim HS, Choi KH. Human mesenchymal stem cells implantation into the degenerated coccygeal disc of the rat. Cytotechnology. 2009 Jan;59(1):55-64. doi: 10.1007/s10616-009-9192-1. Epub 2009 Apr 12. PMID 19363673
- [Background] Hiyama A, Mochida J, Iwashina T, Omi H, Watanabe T, Serigano K, Tamura F, Sakai D. Transplantation of mesenchymal stem cells in a canine disc degeneration model. J Orthop Res. 2008 May;26(5):589-600. doi: 10.1002/jor.20584. PMID 18203202
- [Background] Henriksson HB, Svanvik T, Jonsson M, Hagman M, Horn M, Lindahl A, Brisby H. Transplantation of human mesenchymal stems cells into intervertebral discs in a xenogeneic porcine model. Spine (Phila Pa 1976). 2009 Jan 15;34(2):141-8. doi: 10.1097/BRS.0b013e31818f8c20. PMID 19112334
- [Background] Zhang Y, Drapeau S, Howard SA, Thonar EJ, Anderson DG. Transplantation of goat bone marrow stromal cells to the degenerating intervertebral disc in a goat disc injury model. Spine (Phila Pa 1976). 2011 Mar 1;36(5):372-7. doi: 10.1097/BRS.0b013e3181d10401. PMID 20890267
- [Background] Jeong JH, Lee JH, Jin ES, Min JK, Jeon SR, Choi KH. Regeneration of intervertebral discs in a rat disc degeneration model by implanted adipose-tissue-derived stromal cells. Acta Neurochir (Wien). 2010 Oct;152(10):1771-7. doi: 10.1007/s00701-010-0698-2. Epub 2010 Jun 24. PMID 20571835
- [Background] Chun HJ, Kim YS, Kim BK, Kim EH, Kim JH, Do BR, Hwang SJ, Hwang JY, Lee YK. Transplantation of human adipose-derived stem cells in a rabbit model of traumatic degeneration of lumbar discs. World Neurosurg. 2012 Sep-Oct;78(3-4):364-71. doi: 10.1016/j.wneu.2011.12.084. Epub 2011 Dec 24. PMID 22381275
- [Background] Ganey T, Hutton WC, Moseley T, Hedrick M, Meisel HJ. Intervertebral disc repair using adipose tissue-derived stem and regenerative cells: experiments in a canine model. Spine (Phila Pa 1976). 2009 Oct 1;34(21):2297-304. doi: 10.1097/BRS.0b013e3181a54157. PMID 19934809
- [Background] Miyamoto T, Muneta T, Tabuchi T, Matsumoto K, Saito H, Tsuji K, Sekiya I. Intradiscal transplantation of synovial mesenchymal stem cells prevents intervertebral disc degeneration through suppression of matrix metalloproteinase-related genes in nucleus pulposus cells in rabbits. Arthritis Res Ther. 2010;12(6):R206. doi: 10.1186/ar3182. Epub 2010 Nov 5. PMID 21054867
- [Background] Leckie SK, Sowa GA, Bechara BP, Hartman RA, Coelho JP, Witt WT, Dong QD, Bowman BW, Bell KM, Vo NV, Kramer BC, Kang JD. Injection of human umbilical tissue-derived cells into the nucleus pulposus alters the course of intervertebral disc degeneration in vivo. Spine J. 2013 Mar;13(3):263-72. doi: 10.1016/j.spinee.2012.12.004. Epub 2013 Feb 4. PMID 23384411
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Vadala G, Sowa G, Hubert M, Gilbertson LG, Denaro V, Kang JD. Mesenchymal stem cells injection in degenerated intervertebral disc: cell leakage may induce osteophyte formation. J Tissue Eng Regen Med. 2012 May;6(5):348-55. doi: 10.1002/term.433. Epub 2011 Jun 13. PMID 21671407
- [Background] Hernigou P, Homma Y, Flouzat-Lachaniette CH, Poignard A, Chevallier N, Rouard H. Cancer risk is not increased in patients treated for orthopaedic diseases with autologous bone marrow cell concentrate. J Bone Joint Surg Am. 2013 Dec 18;95(24):2215-21. doi: 10.2106/JBJS.M.00261. PMID 24352775